## Mopsy Research CONSENT FORM

## INFORMED CONSENT FORM \_\_\_\_\_, hereby consent to participate in the research study of "A Comparative Study on Functional Vision in Astigmatic Patients: DAILIES TOTAL1 Toric Contact Lenses vs. Spherical Equivalent Contact Lenses in Asian Eyes". I have read the PATIENT INFORMATION SHEET and INFORMED CONSENT FORM. The study has been explained to me by investigator. I understood all the benefits and the risks associated with this study. I am not giving up any of my legal rights by signing this informed consent form. I have had opportunities to ask questions to investigator and all my questions have been satisfactorily answered. I have received enough information about the study. If the result of my participation in this study caused any physical injury or feel uncomfortable emotionally, the investigator will treat me or refer me for treatment. By signing this informed consent form, I certify that all information provided is true and correct. I consent to participate in this study and understand that I am free to withdraw at any time, without having to give a reason for withdrawing, and the withdrawal will not affect my present and future medical care. I understand that my identity will be kept confidential. I agree to authorize the Research Ethics Committee (REC) and the regulatory authority(ies) a direct access to my original research data for verification of clinical trial procedures and/or data, without violating my confidentiality, to the extent permitted by the applicable laws and regulations. Name of Participant Signature Date (in BLOCK Letter)

I will be given a signed copy of the informed consent form and participant

information sheet for retention.